CLINICAL TRIAL: NCT06185582
Title: Repetitive Applications of Pruritogens and Effects of a Cutaneous-induced Pain Stimulation on Nonhistaminergic Itch Perception
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Silvia Lo Vecchio, Assistant Professor, Aalborg University
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: N-20210046 2nd project
Record Dates: First submitted 2023-11-20; First posted 2023-12-29 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Pain, Burning; Capsaicin
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: The sub-project takes place over three sessions on three consecutive days. The participants will randomly receive two pruritogens and two pain stimulations (heat or capsaicin) in the same and in the opposite arm.
Who Masked: Participant
Masking Description: Participant will be blinded about application of pruritogens.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain (Experimental): A thermode stimulator of 3x3 cm will be placed on the areas and kept in place by means of Velcro tape. The temperature raises 1°C per second from a starting temperature of 32°C until itch reach or 46.5 °C. This temperature will be maintained for 2 minutes. Then the temperature will return to baseline temperature at a rate of 5°C /s.
  Interventions: Other: Cowhage
- Capsaicin (Experimental): Capsaicin patches (dosage form: transdermal patch 8% Qutenza, Astellas) will be applied on one squared area (4x4 cm2). The patch will be left in place for 20 minutes after which it will be removed.
  Interventions: Other: Cowhage

INTERVENTIONS:
Other: Cowhage — 25 spicules will be inserted in the center of the predefined skin area on the mandibular area. The spicules will be gently rubbed for 15-20 seconds in circular motion to facilitate epidermal penetration.

SUMMARY:
In This experiment, the investigators would like to test following hypotheses:

the pain stimulation applied at the same time of a pruriceptive stimulus will decrease the itch perception. Moreover, also the effect of the cutaneous pain stimulus location (same forearm of the pruriceptive stimulus versus the opposite forearm) on histaminergic and non-histaminergic itch will be investigated.

DETAILED DESCRIPTION:
The phenomenon that pain inhibits pain is a well-known mechanism, but it is not known if pain is inhibiting itch. In this context, the aim of this project is to investigate the extent to which thermal or neurogenic short cutaneous pain can affect the itch perception. In particular, the project aims to understand any differences in itch perception when the painful stimulation is applied on the same forearm versus the opposite forearm. The hypothesis is that by applying a painful stimulus at the same time of an itchy stimulus, the itch sensitivity will decrease; probably due to an inhibitory process conducted by interneurons (Bhlbb5 interneuron) at central level.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* 18-60 years
* Speak and understand English

Exclusion Criteria:

* Pregnancy or lactation
* Drug addiction defined as any use of cannabis, opioids, or other addictive drugs
* Previous or current history of neurological (e.g. neuropathy), immunological (e.g. asthma, immune deficiencies, arthritis) musculoskeletal (e.g. muscular pain in the upper extremities,), cardiac disorder, or mental illnesses that may affect the results
* Lack of ability to cooperate
* Current use of medications that may affect the trial such as antihistamines, antipsychotics, and pain killers, as well as systemic or topical steroids
* Skin diseases (e.g. atopic dermatitis, pruritus nodularis, eczema, psoriasis)
* Moles, scars, or tattoos in the area to be treated or tested.
* Consumption of alcohol or painkillers 24 hours before the study days and between these
* Acute or chronic pain
* Participation in other trials within one week of study entry (four weeks in the case of pharmaceutical trials)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of itch intensity using a VAS scale | 1 minute post itch provocation
  Immediately following the itch provocations, participants will be instructed to rate the itch intensity for 10 minutes using a digital visual analogue scale (VAS; eVAS Software: Aalborg, University, Denmark), on a tablet. The scale will be measured from 0 to 100, where 0 represents 'no itch' and 100 'worst itch imaginable'.
Assessment of pain intensity using a VAS scale | 1 minute post itch provocation
  Immediately following the itch provocations, participants will be instructed to rate the pain intensity for 10 minutes using a digital visual analogue scale (VAS; eVAS Software: Aalborg, University, Denmark), on a tablet. The scale will be measured from 0 to 100, where 0 represents 'no pain' and 100 'worst pain imaginable'.
Retrospective rating of the pain perceived on a NRS | 10 minutes post itch provocation
  After 10 minutes of pruritogens application, a retrospective rating of the pain perceived from the thermal pain/capsaicin will be provided by the subject using a numeral rating scale (NRS)

SECONDARY OUTCOMES:
Alloknesis | 12 minutes post itch provocation
  Alloknesis sensation is measured using a standardized sensory brush (SENSELab Brush-05, Somedic AB, Hörby, Sweden) exerting a force of 200 to 400 mN.
Mechanically evoked itch | 15 minutes post itch provocation
  Mechanically evoked itch is measured using three von Frey filaments of 4.08, 4.16 and 4.31 (1.0, 1.4, 2.0 g, respectively) (North Coast Medical, Gilroy, CA). The center of the skin area is stimulated by 3 pricks, repeated 3 times in short succession. After a total of 9 stimulations, the participants will report the itch elicited on a numerical rating scale (NRS) from 0 to 10 (0 = "no itch"; 10 = "worst imaginable itch").

CONTACTS AND LOCATIONS:
Locations (1):
- Aalborg University, Aalborg, Denmark